CLINICAL TRIAL: NCT00001424
Title: Evaluation and Natural History of Children With Cancer and AIDS
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950025; 95-C-0025
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: Acquired Immunodeficiency Syndrome; Cancer; HIV Infections; Leukemia; Lymphoma
Keywords: AIDS; Children; Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Neoplasms; HIV Infections; Leukemia; Lymphoma

SUMMARY:
Patients enrolled in this study will not receive investigational therapy. Any treatments rendered will be standard and based on appropriate medical care. Should a patient become eligible for an experimental therapy protocol, the normal process of enrollment and informed consent will be followed.

DETAILED DESCRIPTION:
This protocol will enable the Pediatric Branch to follow selected children with cancer or HIV infection who are not immediately eligible for protocol enrollment but who are likely, within the next year, to become candidates for protocol entry. It will also enable the Pediatric Branch to follow children who present with either clinical findings that constitute important educational experiences for the NCI trainees or who have unique or unusual medical problems that are likely to benefit from the research expertise of the NCI.

ELIGIBILITY:
Children with cancer (or a precancer syndrome) or HIV infection, between the age(s) of 3 months to 30 years, who are evaluated by the Pediatric Branch and are found to be not immediately eligible for an ongoing protocol but are likely to become a candidate for a future protocol.

Children with cancer (or a precancer syndrome) or HIV infection, who present with disease manifestations of special interest to Pediatric Branch investigators, because they are likely to shed light on disease.

Patients who, when evaluated by the Branch, are determined to likely never become eligible for a Pediatric Branch protocol are not eligible for this protocol.

No patients younger than 3 months of age or older than 30 years of age are eligible for this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110
Dates: Start 1994-11; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States